CLINICAL TRIAL: NCT01909310
Title: Head Positions to Open the Upper Airway IV
Brief Title: Head Positions to Open the Airway IV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Principal Investigator, Peter Paal, PD MD MBA EDAIC EDIC, PD Dr. Peter Paal, EDAIC, EDIC, Medical University Innsbruck
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UN5155 327/4.10
Record Dates: First submitted 2013-07-24; First posted 2013-07-26 (Estimated); Last update posted 2017-03-23 (Actual); Status verified 2017-03

CONDITIONS: Cardiac or Respiratory Arrest, Anaesthesia
Keywords: anesthesia, cardiac arrest, resuscitation, ventilation
MeSH Terms: conditions — Apnea; Heart Arrest; Respiratory Aspiration

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- with head support (Active Comparator): patients are ventilated with their heads positioned on a support
  Interventions: Procedure: head extension; Procedure: neutral position; Procedure: anaesthesiologist´s position
- without head support (Sham Comparator): patients are ventilated without head support
  Interventions: Procedure: head extension; Procedure: neutral position; Procedure: anaesthesiologist´s position

INTERVENTIONS:
Procedure: head extension — the lungs are ventilated with the patient´s head extended
Procedure: neutral position — the lungs are ventilated with the patient´s head in neutral position
Procedure: anaesthesiologist´s position — the lungs are ventilated with the patient´s head positioned deemed ideal by the anaesthesiologist

SUMMARY:
After routine induction of general anaesthesia peak airway pressure (= P max) and other respiratory parameters(i.e. expiratory tidal volume, expiratory CO2) are measured with and without head support in three different head positions: neutral position, reclination of the head, a position deemed ideal by the anaesthesist; primary study goal is pmax depending on different head positions;

ELIGIBILITY:
Inclusion Criteria:

* male and female patients ≥ 18 years
* elective operations in general anaesthesia
* patient´s written informed consent
* American Society of Anesthesiology scale I-III

Exclusion Criteria:

* non fasting patient
* body mass index > 35 kg/m2
* anamnestic cervical spine pathologies or other peripheral neurological deficiences due to pathologies of the cervical spine
* malformations of the head or upper airway
* history of perforation of stomach or esophagus
* anamnestic hiatus hernia or reflux
* acute respiratory infection or obstructive airway disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2013-09; Primary Completion 2014-04 (Actual); Study Completion 2015-04-01 (Actual)

PRIMARY OUTCOMES:
Peak airway pressure | peak airway pressure is measured over one minute

CONTACTS AND LOCATIONS:
Locations (1):
- Klinik für Anästhesie und Allgemeine Intensivmedizin, Medizinische Universität Innsbruck, Anichstraße 35, Innsbruck, Austria